CLINICAL TRIAL: NCT04046068
Title: Improving Patient Outcomes Using Multimodal Perioperative Pain Management: The ComfortSafe Program
Brief Title: Multimodal Perioperative Pain Management: ComfortSafe Program
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Georgetown University (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-0854
Record Dates: First submitted 2019-07-17; First posted 2019-08-06 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Post-operative Pain; Post-operative Nausea and Vomiting; Respiratory Depression; Confusion Postoperative
MeSH Terms: conditions — Pain, Postoperative; Vomiting; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: ComfortSafe Care — In most cases, sevoflurane, an inhalation anesthetic, will be used in higher-than-traditional concentrations to replace opioids and provide safe control of vital signs along with amnesia and analgesia. Intravenous (IV) propofol, esmolol, and other beta-blockers can also be administered to prevent increases in BP and HR during surgery. At the time of wound closure, the ComfortSafe Pyramid derived Preemergence Analgesic Checklist guides the anesthesia and surgical teams through collaborative decisions for implementation of a multimodal analgesic plan. Local anesthetics, including liposomal bupivacaine, can then be injected and IV non-opioid analgesics administered allowing the patient to awaken comfortably from anesthesia. Standardized kits for liposomal bupivacaine administration will be utilized. If the patient does have pain, IV opioids can be administered to provide immediate relief without hesitation since the non-opioid analgesics have already been given.

SUMMARY:
Proposed is a demonstration project to characterize the immediate, short-term and long-term pain and other post-operative outcomes of 60, self-selected breast (n=20), caesarian-section (n=20) and abdominal (n=20) surgical patients who receive opioid-sparing, multimodal anesthesia and pain management care as guided by the ComfortSafe Pyramid.

DETAILED DESCRIPTION:
In well-characterized samples of patients undergoing breast, caesarian-section or abdominal surgery, the efficacy and safety of perioperative pain care organized by ComfortSafe Pyramid approaches will be evaluated. In addition, patient satisfaction with this care will be evaluated. Post-operative pain and opioid-related outcomes will be operationalized using standardized symptom (nausea, vomiting, respiratory depression, confusion, acute and chronic pain) severity measures, prn analgesic (opioid and non-opioid) consumption, and urine toxicology. Together, these original data will have important implications for the clinical management of post-operative pain utilizing opioid-sparing and multi-modal approaches.

A total of 60 self-selected surgical patients will be enrolled in the study, 20 undergoing breast surgery, 20 undergoing caesarian-section, and 20 undergoing abdominal surgery. All will receive anesthesia and pain management consistent with the ComfortSafe Pyramid which emphasizes opioid-sparing and multimodal approaches. Side and adverse opioid-related effects and post-operative pain will be assessed at regular intervals during the immediate post-operative period (24 hours). To evaluate the incidence of opioid misuse/abuse and the development of chronic pain, an opioid use history, urine toxicology and Brief Pain Inventory will be collected at 1 month, 3 months and 6 months following discharge. Patient satisfaction measures will be obtained at discharge, 1 month, and 3 months follow-up timepoint.

ELIGIBILITY:
Inclusion Criteria:

1. Be between the ages of 21 and 75 years of age.
2. Be eligible to receive bupivacaine liposomal injectable suspension.
3. Be undergoing a planned inpatient surgical (breast, caesarian-section or abdominal) procedure with general anesthesia.
4. Provide an opioid-free urine prior to surgical procedure.
5. Have a supportive, significant other willing to facilitate patient adherence to ComfortSafe program
6. Be agreeable to study procedures and capable of signing an informed consent.

Exclusion Criteria:

1. Be on chronic opioid therapy for chronic pain or treatment of opioid use disorder.
2. Have chronic pain.
3. Have an active substance use disorder on alcohol, benzodiazepine, methamphetamine, cocaine or other drugs of abuse (except nicotine).
4. Be acutely psychotic, severely depressed and in need of inpatient treatment, or an immediate suicide risk.
5. Have a neurological or psychiatric illness (i.e., schizophrenia, quadriplegia, stroke) that would affect pain responses.
6. Be undergoing a surgical procedure for which liposomal bupivacaine cannot be used (eg. Skin graft, wound debridement, ureteroscopy, hysteroscopy, eye surgery).
7. Have a diagnosis of Obstructive Sleep Apnea with use of CPAP
8. Have an ASA score of 2 or greater as determined by the anesthesiologist.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients preparing to undergo surgery will be recruited from the Pre-Anesthesia Testing (PAT) unit in the Department of Anesthesiology at Medstar Georgetown University Hospital (MGUH). The staff nurse practitioner will inform all patients scheduled for caesarian-section or abdominal surgery of the ComfortSafe program, and provide them a patient education brochure for their review. If a patient is interested in participating in the program, he or she will be instructed to contact the study research nurse to learn more about participation and consider enrolling. Subjects will therefore be self-selected and enrolled on a rolling, convenience basis.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-05-11 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Post-operative Pain: VAS | 24 hours
  Severity of post-operative pain will be operationalized as both (1) responses on a visual analogue pain scale (VAS) and (2) consumption of analgesic medications. The VAS ranges from 0 (no pain) to 10 (worst pain imaginable). Dose and type of analgesic medications consumed during the first 24 hours postoperatively will be abstracted from the electronic record and total amount of each entered into the study database. Opioids administered will be converted into morphine equivalent doses (MED) for analysis.
Post-operative nausea and vomiting | 24 hours
  The incidence and severity of post-operative nausea and vomiting experienced by the subjects will be measured at each time point using Postoperative Nausea and Vomiting (PONV) impact scale. This tool records the frequency, intensity and duration of nausea, as well as the number of vomits, and designed to detect minimal clinically important differences. Specifically, the tool uses ordinal responses to quantify nausea intensity and impact on the patient, where (i)=0, (ii)=1, (iii)=2, and (iv)=3. In addition, the number of vomits are used to quantify vomiting intensity, scored as the number of vomits (0-2, or 3 if three or more vomits); both scores are added together to obtain the simplified PONV impact scale score. When anitemetics are used, their dose and timing will be recorded.
respiratory depression | 24 hours
  Respiratory depression will be scored as present (respiratory rate ≤ 10 breaths/minute) or absent (respiratory rate > 10 breaths/minute)
confusion post-operative | 24 hours
  Post-operative confusion will be assessed with the Delirium Observation Screening (DOS) scale, a 13-item scale developed to facilitate early recognition of delirium according to Diagnostic and Statistical Manual-IV criteria. Evaluated on a 4pt Likert scale (0-never, 4-always) are, consciousness; attention; thinking; memory; psychomotor activity; sleep/wake; mood; and perception, with items totaled to provide an overall delirium score. The scale boasts good internal consistency, and content, predictive, concurrent and construct validity in adult and elderly populations.

SECONDARY OUTCOMES:
Chronic Post-surgical Pain | 1 month, 3 months and 6 months
  To capture the presence and severity of ongoing pain, the Brief Pain Inventory (BPI) will be administered. This tool goes beyond measurement of the intensity of pain (sensory dimension), to evaluate interference by pain in the patient's life (reactive dimension), as well as pain relief, pain quality, and the patient's perception of the cause of pain. With respect to functionality, the BPI asks for ratings of the degree to which pain interferes with mood, walking and other physical activity, work, social activity, relations with others, and sleep; using numeric 0 to 10 scales, with 0 being "no interference" and 10 being "interferes completely," the mean of these scores is used as a pain interference score. For analysis, the pain worst rating can be chosen to be the primary response variable, with the other items serving as a check on variability, or, alternatively, the ratings can be combined to give a composite index of pain severity.
Chronic Post-surgical opioid consumption | 1 month, 3 months and 6 months
  Patients will be discharged with an analgesic use diary and daily MME will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Medstar Georgetown University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No